CLINICAL TRIAL: NCT02830113
Title: Effects of Non-surgical Treatment of Chronic Periodontitis on Insulin Resistance and Glucose Tolerance in Non-diabetic Subjects
Brief Title: Metabolic Effects of Treatment of Chronic Periodontitis in Non-diabetic Subjects
Acronym: PARODIA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Professor of Endocrinology and Diabetes, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CNO20155
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Periodontitis; Prediabetes
Keywords: periodontitis; diabetes; prevention; impaired glucose tolerance; insulin resistance
MeSH Terms: conditions — Periodontitis; Prediabetic State; Diabetes Mellitus; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-surgical periodontal treatment (Experimental): One session of non-surgical periodontal treatment consisting of a complete scaling, polishing, root planning, and the irrigation of periodontal pockets with a 10% povidone iodine solution.
  Interventions: Procedure: non-surgical periodontal treatment

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — One session of complete scaling, polishing, root planning, and the irrigation of periodontal pockets with a 10% povidone iodine solution

SUMMARY:
This study was aimed at assessing the effects of non-surgical periodontal treatment (NSPT) of chronic periodontitis on insulin sensitivity, glucose tolerance, and serum C-reactive protein(CRP) level amongst non-diabetic subjects.

DETAILED DESCRIPTION:
Subjects with chronic periodontitis will undergo non-surgical periodontal treatment (NSPT) consisting of a complete scaling, polishing, root planning, and the irrigation of periodontal pockets with a 10% povidone iodine solution. Periodontal parameters (plaque index, gingival bleeding index, pocket depth, and clinical attachment loss), insulin sensitivity using KITT, glucose tolerance using oral glucose tolerance test and serum CRP level by immunoturbidimetry will be measured before and 3 months after the NSPT.

ELIGIBILITY:
Inclusion Criteria:

* Chronic periodontitis
* Non diabetic individual

Exclusion Criteria:

* Known diabetes
* Periodontal treatment less than 6 months prior to inclusion
* Having less than 20 natural teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 3 months
  change in 2-hour post load blood glucose
Insulin sensitivity | 3 months
  change in glucose disappearance rate during the short insulin tolerance test

SECONDARY OUTCOMES:
Composite periodontal health | 3 months
  Change in plaque index, gingival bleeding index, pocket depth, and clinical attachment loss
Inflammation | 3 months
  change in Serum CRP

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobngwi, MD, PhD, Principal Investigator — University of Yaoundé 1 and Yaoundé Central Hospital

REFERENCES:
- [Derived] Nana Nana AR, Tsobgny Tsague NF, Lontchi-Yimagou E, Bengondo Messanga C, Tankeu A, Katte JC, Balti Vounsia E, Dehayem M, Sobngwi E. Effects of non-surgical treatment of chronic periodontitis on insulin resistance and glucose tolerance in subjects without diabetes (PARODIA 2 study). J Investig Med. 2021 Oct;69(7):1377-1381. doi: 10.1136/jim-2021-001831. Epub 2021 Jul 14. PMID 34261767